CLINICAL TRIAL: NCT06554535
Title: A Single-center, Single-arm, Prospective Clinical Study to Evaluate the Efficacy and Safety of Serplulimab in Combination With Platinum-based Chemotherapy and Bayer Aspirin in Previously Untreated Patients With Extensive-stage Small Cell Lung Cancer.
Brief Title: Efficacy and Safety of Serplulimab With Chemotherapy and Aspirin in Untreated Extensive-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB20240810
Record Dates: First submitted 2024-08-10; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Extensive-Stage Small Cell Lung Cancer; Treatment-naïve for Systemic Therapy Targeting Extensive-Stage Small Cell Lung Cancer; ECOG Performance Status Score of 0 or 1; Expected Survival ≥3 Months
Keywords: ES-SCLC; Chemo-immunotherapy combination; Aspirin
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab + Chemotherapy + Aspirin (Experimental)
  Interventions: Drug: Serplulimab，Platinum-based Chemotherapy，Aspirin

INTERVENTIONS:
Drug: Serplulimab，Platinum-based Chemotherapy，Aspirin — Participants will receive an induction therapy consisting of Serplulimab (4.5 mg/kg IV on Day 1), Carboplatin (AUC 5 IV on Day 1) or Cisplatin (75 mg/m² IV on Day 1), Etoposide (100 mg/m² IV on Days 1-3), and Bayer Aspirin (100 mg PO daily). This induction phase will be administered every 3 weeks for 4 cycles. Following the induction phase, participants will transition to a maintenance therapy phase where they will continue to receive Serplulimab (4.5 mg/kg IV on Day 1, every 3 weeks) and Bayer Aspirin (100 mg PO daily) until disease progression or intolerable toxicity.

SUMMARY:
Lung cancer remains a leading cause of cancer-related deaths worldwide, with small cell lung cancer (SCLC) accounting for 15-20% of all lung cancers. Extensive-stage SCLC (ES-SCLC) is associated with poor prognosis, with a median survival of 2-4 months without treatment. Although platinum-based chemotherapy is the standard first-line treatment, median survival remains under one year, highlighting the need for improved outcomes. Recent studies have demonstrated that combining PD-1 inhibitors with chemotherapy can significantly improve survival in ES-SCLC patients. Serplulimab, a novel PD-1 inhibitor, has shown promising results in extending overall survival when combined with chemotherapy in a Phase III trial. Additionally, aspirin has been found to enhance the anti-tumor effects of immunotherapy by inhibiting immune checkpoint proteins and reducing adverse events such as thrombosis and fever. This Phase II study aims to evaluate the efficacy and safety of combining serplulimab, platinum-based chemotherapy, and aspirin as a first-line treatment for patients with ES-SCLC.

DETAILED DESCRIPTION:
In 2020, global cancer burden data showed 2.2 million new cases of lung cancer, ranking second, with 1.8 million deaths, far surpassing other cancer types and ranking first in cancer-related mortality. In 2020, China reported 820,000 new cases of lung cancer, with 710,000 deaths, accounting for 23.8% of all cancer deaths, making lung cancer the leading cause of cancer incidence and mortality in the country. Small cell lung cancer (SCLC), originating from neuroendocrine-differentiated epithelial cells, accounts for 15-20% of all lung cancers. Using the Veterans Administration (VA) staging system, SCLC is classified into limited-stage and extensive-stage disease. The majority of patients present with symptoms related to metastatic lesions at diagnosis, and only 30-40% are diagnosed at the limited stage. Extensive-stage patients, due to widespread metastasis and poor physical condition, often can only receive supportive care, resulting in shorter survival times.

Based on theoretical foundations, cytotoxic chemotherapy kills tumor cells (TC), exposing the immune system to high levels of tumor antigens. Therefore, compared to standard chemotherapy alone, activating tumor-specific T-cell immunity by inhibiting the PD-L1/PD-1 signaling pathway may provide deeper and more durable responses. Recent studies have explored the potential of combining immunotherapy with chemotherapy as a first-line treatment for extensive-stage small cell lung cancer (ES-SCLC).

Serplulimab is an innovative PD-1 inhibitor developed by Henlius, a recombinant humanized IgG4 monoclonal antibody. It has characteristics such as structural stability, weak antibody-dependent cellular cytotoxicity (ADCC) and complement-dependent cytotoxicity (CDC), moderate antibody-dependent cellular phagocytosis (ADCP) effects, large epitope binding area, high affinity, slow dissociation, strong anti-tumor activity, and low immunogenicity. Clinical studies involving serplulimab combined with chemotherapy as a first-line treatment for extensive-stage small cell lung cancer have been conducted to evaluate its safety and efficacy.

Aspirin (ASP), originally extracted from willow bark, is a small molecule compound with various effects such as antipyretic, anti-inflammatory, analgesic, and antiplatelet aggregation. In recent years, research has discovered new anti-cancer effects of aspirin, and it has been confirmed to promote tumor cell apoptosis. Additionally, preclinical evidence suggests that antiplatelet drugs and immune checkpoint inhibitors (ICIs) may have potential synergistic effects, which warrant further investigation in the context of lung cancer treatment.

PD-1 inhibitors, as the standard first-line treatment for extensive-stage small cell lung cancer, have been proven in numerous studies to have good efficacy and safety. Aspirin, as a classic anticoagulant, has advantages such as safety, affordability, and easy availability. Lung cancer patients are inherently in a hypercoagulable state, and if aspirin's synergistic anti-tumor effects and its potential to reduce adverse events such as fever and thrombosis can be further confirmed, it will have a significant impact on the treatment of ES-SCLC patients, potentially achieving enhanced therapeutic effects. Therefore, we plan to conduct this observational Phase II study to evaluate the efficacy and safety of combining the PD-1 inhibitor serplulimab, platinum-based chemotherapy, and Bayer aspirin as first-line treatment for extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years.
2. Histologically or cytologically confirmed ES-SCLC (according to the Veterans Administration Lung Cancer Group [VALG] staging system).
3. Treatment-naïve for systemic therapy targeting ES-SCLC.
4. Patients must have at least one tumor lesion that meets the following criteria: previously untreated, accurately measurable, with a longest diameter ≥ 10 mm at baseline (for lymph nodes, short axis ≥ 15 mm), measurable by chest CT or PET-CT, as long as accurate repeat measurements can be performed.
5. ECOG performance status score of 0 or 1.
6. Expected survival ≥ 3 months.
7. Planned treatment with Serplulimab combined with platinum-based chemotherapy.
8. Patients who have previously taken or are currently taking Bayer Aspirin are allowed.

Exclusion Criteria:

1. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.
2. Currently receiving other anticoagulant therapy.
3. Previous systemic anti-tumor therapy.
4. Contraindications to the use of Serplulimab, Aspirin, or chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Up to 2 years
  The time from the start of treatment until the first documented disease progression or death from any cause, whichever occurs first, as assessed by RECIST criteria (Response Evaluation Criteria in Solid Tumors).

SECONDARY OUTCOMES:
Two-Year Overall Survival | 2 years
  The proportion of patients still alive two years after the start of treatment.
Objective Response Rate | Up to 2 years
  The proportion of patients with a measurable reduction in tumor size as per RECIST criteria, including complete and partial responses.
Disease Control Rate | Up to 2 years
  The proportion of patients who achieve complete response (CR), partial response (PR), or stable disease (SD) as per RECIST criteria.
Incidence of Adverse Events | Up to 2 years
  The number and severity of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheng Y, Han L, Wu L, Chen J, Sun H, Wen G, Ji Y, Dvorkin M, Shi J, Pan Z, Shi J, Wang X, Bai Y, Melkadze T, Pan Y, Min X, Viguro M, Li X, Zhao Y, Yang J, Makharadze T, Arkania E, Kang W, Wang Q, Zhu J; ASTRUM-005 Study Group. Effect of First-Line Serplulimab vs Placebo Added to Chemotherapy on Survival in Patients With Extensive-Stage Small Cell Lung Cancer: The ASTRUM-005 Randomized Clinical Trial. JAMA. 2022 Sep 27;328(12):1223-1232. doi: 10.1001/jama.2022.16464. PMID 36166026